CLINICAL TRIAL: NCT00605293
Title: An Open Label Randomised Controlled Study to Compare the Efficacy, Safety and Tolerability of Once-monthly Administration of Intravenous C.E.R.A. Versus Epoetin Alfa for the Maintenance of Haemoglobin Levels in Hemodialysis Patients With Chronic Renal Anaemia
Brief Title: A Study of Intravenous Mircera (C.E.R.A or Methoxy Polyethylene Glycol-epoetin Beta) for the Maintenance Treatment of Hemodialysis Participants With Chronic Renal Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML21060; 2007-002065-12 (EudraCT Number)
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Results first posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2013-10

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator; Epoetin Alfa

ARMS (2):
- C.E.R.A (Experimental): Participants received starting dose of 120, 200 or 360 mcg of C.E.R.A IV once monthly for 6 months. The starting dose was based on the dose of epoetin alfa administered in Week -1.
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta
- Epoetin Alfa (Active Comparator): Participants received IV injection of 6000 International Units (IU) of epoetin alfa every 3 weeks (q3wk) during the Stability Verification Period (SVP; Week -4 to -1), and 7443 IU of epoetin alfa q3wk during Dose Titration Period (DTP; Week 0 to 15), 7363 IU of epoetin alfa q3wk during Efficacy Evaluation Period (EEP; Week 16 to 23) up to 23 weeks.
  Interventions: Drug: Epoetin alfa

INTERVENTIONS:
Drug: methoxy polyethylene glycol-epoetin beta — 120, 200 or 360 micrograms iv/month (starting dose)
  Other Names: Mircera; C.E.R.A
  Arms: C.E.R.A
Drug: Epoetin alfa — As prescribed
  Arms: Epoetin Alfa

SUMMARY:
This 2 arm study will compare the efficacy and safety of monthly administration of intravenous (IV) Mircera versus epoetin alfa for the maintenance of hemoglobin levels in hemodialysis patients with chronic renal anemia. Participants currently receiving maintenance treatment with epoetin alfa will be randomized either to receive monthly injections of 120, 200 or 360 micrograms Mircera, with the starting dose derived from the dose of epoetin alfa they were receiving in the week preceding study start, or to continue on epoetin alfa treatment. The anticipated duration of study is 32 weeks, and the target sample size is 146 participants.

ELIGIBILITY:
Inclusion Criteria:

* chronic renal anemia;
* continuous iv maintenance epoetin alfa therapy, with the same dosing interval during the previous month to and during SVP;
* regular hemodialysis for greater than or equal to (>=) 3 months

Exclusion Criteria:

* transfusion of red blood cells during previous 2 months
* poorly controlled hypertension requiring interruption of epoetin alfa treatment in previous 6 months;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2008-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (16):
- Spain (16):
  - Badajoz, Badajoz
  - Barcelona, Barcelona
  - Cáceres, Caceres
  - Cádizv, Cadiz
  - Castellon, Castellon
  - Ciudad Real, Ciudad Real
  - Huelva, Huelva
  - Madrid, Madrid
  - Marbella, Malaga
  - Tudela, Navarre
  - Pontevedra, Pontevedra
  - Salamanca, Salamanca
  - Teruel, Teruel
  - Valencia, Valencia
  - Zamora, Zamora
  - Zaragoza, Zaragoza

REFERENCES:
- [Derived] Locatelli F, Choukroun G, Truman M, Wiggenhauser A, Fliser D. Once-Monthly Continuous Erythropoietin Receptor Activator (C.E.R.A.) in Patients with Hemodialysis-Dependent Chronic Kidney Disease: Pooled Data from Phase III Trials. Adv Ther. 2016 Apr;33(4):610-25. doi: 10.1007/s12325-016-0309-6. Epub 2016 Mar 10. PMID 26965694

RESULTS

PARTICIPANT FLOW:
Groups:
- C.E.R.A: Participants received starting dose of 120, 200 or 360 micrograms (mcg) of C.E.R.A intravenously (IV) once monthly for 6 months. The starting dose was based on the dose of epoetin alfa administered in Week -1.
- Epoetin Alfa: Participants received IV injection of 6000 International Units (IU) of epoetin alfa every 3 weeks (q3wk) during the Stability Verification Period (SVP; Week -4 to -1), 7443 IU of epoetin alfa q3wk during Dose Titration Period (DTP; Week 0 to 15), and 7363 IU of epoetin alfa q3wk during Efficacy Evaluation Period (EEP; Week 16 to 23) up to 23 weeks.
Period: Overall Study
Arm/Group | C.E.R.A | Epoetin Alfa
Started | 65 | 36
Completed | 48 | 31
Not Completed | 17 | 5
Not completed — Death | 2 | 1
Not completed — Insufficient Therapeutic Response | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Holidays Dialysis Out | 1 | 0
Not completed — Blood Transfusion | 7 | 1
Not completed — Renal Transplantation | 3 | 1
Not completed — Incorrect Epoetin Beta Administration | 1 | 0
Not completed — Dialysis Out of Centre for 3 Months | 0 | 1
Not completed — Principal Investigator Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who received at least one dose of C.E.R.A. or epoetin alfa after Week 0, and for whom, data for at least one follow-up variable was available.
Groups:
- Epoetin Alfa: Participants received IV injection of 6000 IU of epoetin alfa q3wk during the SVP (Week -4 to -1), 7443 IU of epoetin alfa q3wk during DTP (Week 0 to 15), and 7363 IU of epoetin alfa q3wk during EEP (Week 16 to 23) up to 23 weeks.
- Total: Total of all reporting groups
Arm/Group | C.E.R.A | Epoetin Alfa | Total
Number analyzed (Participants) | 65 | 36 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (14.93) | 64.5 (16.62) | 64.9 (15.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 17 | 46
  Male | 36 | 19 | 55

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Maintained Average Hemoglobin (Hb) Concentration Within Plus Minus (+/-) 1 Grams Per Deciliter (g/dL) of Their Reference Hb and Between 10 and 12 g/dL During the EEP
Description: Participants who maintained average Hb concentration within +/-1 g/dL of their reference Hb and between 10 to 12 g/dL during EEP are reported. The reference Hb value was defined on the basis of all assessments at Weeks -4, -3, -2, -1 and 0.
Time Frame: EEP (Week 16 to 23)
Population: Per Protocol (PP) population was as a subset of the ITT population who completed the study without any major protocol deviations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C.E.R.A | Epoetin Alfa
Number analyzed (Participants) | 44 | 29
percentage of participants | 45.45 [30.39 to 61.15] | 55.17 [35.69 to 73.55]
Statistical Analysis 1: Comparison: C.E.R.A vs Epoetin Alfa; Test type: Superiority or Other; p = 0.4778, Fisher Exact

2. Secondary Outcome: Change in Hb Concentrations Between Baseline SVP and the EEP
Description: Change in Hb concentration between baseline SVP and the EEP was evaluated by subtracting the mean of Hb concentration during the SVP (Weeks -4 to -1) with the mean of Hb concentration during the EEP (Weeks 16 to 23).
Time Frame: SVP (Week -4 to -1), EEP (Week 16 to 23)
Population: ITT population.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | C.E.R.A | Epoetin Alfa
Number analyzed (Participants) | 65 | 36
g/dL | -0.35 (1.32) | 0.32 (1.06)

3. Secondary Outcome: Percentage of Participants Who Maintained Hb Concentration Between 10 and 12 g/dL Throughout the EEP
Description: Participants who maintained Hb concentration between 10 to 12 g/dL throughout the EEP are reported.
Time Frame: EEP (Week 16 to 23)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | C.E.R.A | Epoetin Alfa
Number analyzed (Participants) | 65 | 36
percentage of participants | 32.7 | 40.6

4. Secondary Outcome: Mean Time Spent in Hb Range 10-12 g/dL
Time Frame: SVP (Week -4 to -1), DTP (Week 0 to 15), and EEP (Week 16 to 23)
Population: ITT population. Here, n = participants who were evaluable for each category, for respective arm groups.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | C.E.R.A | Epoetin Alfa
Number analyzed (Participants) | 65 | 36
days
  SVP (Week -4 to -1) (n=65, 36) | 26.7 (4.46) | 27.1 (4.74)
  DTP (Week 0 to 15) (n=65, 36) | 67.5 (33.92) | 72.9 (37.03)
  EEP (Week 16 to 23) (n=55, 32) | 32.2 (18.25) | 28.9 (21.53)

5. Secondary Outcome: Percentage of Participants Who Required Dose Adjustments During the DTP and EEP
Time Frame: DTP (Week 0 to 15) and EEP (Week 16 to 23)
Population: Safety population included all those participants who were treated with at least one dose of the trial medication and had a safety follow-up, whether withdrawn prematurely or not. Here, "n" = participants who were evaluable for each category, for respective arm groups.
Measure: Number; unit: percentage of participants
Arm/Group | C.E.R.A | Epoetin Alfa
Number analyzed (Participants) | 65 | 36
percentage of participants
  DTP: No dose change (n=65, 36) | 30.8 | 44.4
  DTP: Any dose change (n=65, 36) | 67.7 | 55.6
  DTP: Dose increased (n=65, 36) | 18.5 | 19.4
  DTP: Dose decreased (n=65, 36) | 24.6 | 25.0
  DTP: Dose decreased and increased (n=65, 36) | 24.6 | 11.1
  DTP:Only one dose changed (n=65,36) | 1.5 | 0.0
  EEP: No dose change (n=55, 32) | 60.0 | 65.6
  EEP: Any dose change (n=55, 32) | 30.9 | 34.4
  EEP: Dose increased (n=55, 32) | 20.0 | 12.5
  EEP: Dose decreased (n=55, 32) | 10.9 | 18.8
  EEP: Dose decreased and increased (n=55, 32) | 0.0 | 3.1
  EEP: Only one dose changed (n=55, 32) | 9.1 | 0.0

6. Secondary Outcome: Percentage of Participants Who Received Red Blood Cell (RBC) Transfusions During DTP and EEP
Description: RBC transfusions could be given during the study in case of medical need, i.e., in severely anemic participants with recognized symptoms or signs of anemia (e.g., in participants with acute blood loss, with severe angina, or whose hemoglobin decreased to critical levels).
Time Frame: DTP (Week 0 to 15) up to EEP (Week 16 to 23)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | C.E.R.A | Epoetin Alfa
Number analyzed (Participants) | 65 | 36
percentage of participants | 12.3 | 2.8

ADVERSE EVENTS:
Time Frame: Week 0 to Week 28
Arm/Group | C.E.R.A | Epoetin Alfa
Serious Adverse Events (participants affected / at risk) | 16/65 | 4/36
Other Adverse Events (participants affected / at risk) | 11/65 | 9/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | C.E.R.A (N=65) | Epoetin Alfa (N=36)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Bronchiectasis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Lung infection pseudomonal (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Ischaemic neuropathy (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | C.E.R.A (N=65) | Epoetin Alfa (N=36)
Atrial fibrillation (Cardiac disorders) | 5 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 2
Hypertension (Vascular disorders) | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.